CLINICAL TRIAL: NCT05978102
Title: An Open-label, Dose Escalation and Dose Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of STI-7349 in Subjects With Advanced Solid Tumors
Brief Title: A Dose Escalation and Dose Expansion Clinical Study of STI-7349 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2023-092
Record Dates: First submitted 2023-06-25; First posted 2023-08-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab; spartalizumab; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STI-7349 alone (Experimental): Dose escalation and dose expansion for STI-7349 alone,to determine the RP2D and to evaluate the preliminary antitumor activity of STI-7349 in specific solid tumor patients.
  Interventions: Drug: STI-7349
- STl-7349 in combination with Pembrolizumab (Experimental): Dose escalation and dose expansion for STI-7349 in combination with Pembrolizumab,to determine the RP2D of STI-7349 in combination with Pembrolizumab and to evaluate the preliminary antitumor activity in specific solid tumor patients.
  Interventions: Drug: STI-7349; Drug: Pembrolizumab; Drug: Standard treatment（SoC）
- STl-7349 in combination with other approved PD-1/PD-L1 inhibitors (Experimental): Dose escalation and dose expansion for STI-7349 in combination with with other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.), to determine the RP2D of STI-7349 in combination with Pembrolizumab and to evaluate the preliminary antitumor activity in specific solid tumor patients.
  Interventions: Drug: STI-7349; Drug: Standard treatment（SoC）; Drug: approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.)

INTERVENTIONS:
Drug: STI-7349 — Administered by intravenous infusion (IV)
  Other Names: IL2v mRNA
Drug: Pembrolizumab — Administered by intravenous infusion (IV)
  Other Names: anti-PD-1 monoclonal antibody
  Arms: STl-7349 in combination with Pembrolizumab
Drug: Standard treatment（SoC） — Depending on the treatment stage of enrolled subjects, the investigator will determine the standard treatment regimen and dosage with reference to the CSCO or other current guidelines.
  Other Names: Standard treatment
  Arms: STl-7349 in combination with Pembrolizumab; STl-7349 in combination with other approved PD-1/PD-L1 inhibitors
Drug: approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) — Depending on the treatment stage of enrolled subjects, the investigator will determine the standard treatment regimen and dosage with reference to the CSCO or other current guidelines or the corresponding drug Labeling.
  Arms: STl-7349 in combination with other approved PD-1/PD-L1 inhibitors

SUMMARY:
This is a first-in-human, Phase Ⅰ, open-label, 2-period dose escalation and expansion study of STI-7349 administered intravenously to subjects with advanced solid tumors:

* Period I is divided into two parts: Dose escalation for STI-7349 alone (1A) and dose expansion for STI-7349 alone (1B). In Part 1A, a rapid titration approach and traditional 3 + 3 trial design will be used to assess the safety, dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), PK/biomarker profile, and to determine the recommended Phase 2 dose (RP2D) of STI-7349 alone; in Part 1B, an expansion study of STI-7349 alone will be conducted in target tumor types that may potentially benefit to assess the safety and preliminary efficacy of STI-7349 alone.
* Period Ⅱ is divided into two parts: Dose escalation for STI-7349 in combination with Pembrolizumab (2A) or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) and dose expansion for STI-7349 in combination with Pembrolizumab (2B) or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.). In Part 2A, a dose escalation study of STI-7349 in combination with Pembrolizumab or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) is planned to be conducted using ½ RP2D of STI-7349 alone as the starting dose, which will use a traditional 3 + 3 trial design to assess the safety, DLTs, MTD, PK/biomarker profile of STI-7349 in combination with Pembrolizumab or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) , and to determine the RP2D of STI-7349 in combination with Pembrolizumab or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) ; in Part 2B, an expansion study of STI-7349 in combination with Pembrolizumab or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) or add standard treatment on the basis of STI-7349 combined with pembrolizumab or Other approved PD-1/PD-L1 inhibitors on the market (such as tislelizumab, etc.) will be conducted in target tumor types that may potentially benefit to assess the safety and preliminary efficacy of the combination.

DETAILED DESCRIPTION:
Period I: Dose escalation of STI-7349 alone (1A) Periond 1A1 part: According to the preclinical trial data, 1mg was used as the initial dose and the accelerated titration test design was adopted. If no adverse events have occurred as specified in the following acceleration titers, the dose increment ratio of 60%, 50%, 50%, 33.3%, 25% is recommended by the modified Fibonacci method. The six initial dose groups of STI-7349 were 1mg, 1.6mg, 2.4mg, 3.6mg, 4.8mg and 6.0 mg.respectively. Eligible subjects will be placed into 6 dose groups in sequence from low to high dose.

Subjects in all dose groups will receive 21 days per dosing cycle and Day 1 of each cycle will be the dosing day.

Part 1A1 of this trial will use rapid titration and a traditional 3 + 3 trial design.

Periond 1A2 part: According to the preliminary clinical trial data available , the terminal elimination half-life of HSA-IL2v in humans is approximately 23 hours. With reference to the modified Fibonacci method, the dose escalation ratio is set at 60%. Therefore, two preliminary dose levels for STI-7349 escalation have been established: 1 mg and 1.6 mg. Eligible subjects will be sequentially enrolled into the two dose groups in ascending order.

For all dose groups, each treatment cycle will last 28 days, with dosing administered on Day 1 and Day 15 of each cycle.

The Part 1A2 of this trial will adopt the conventional "3+3" study design. Period I: Dose expansion of STI-7349 alone (1B) Based on data from the 1A escalation period, target tumor types with potential benefit are selected, and subjects are expanded to 20 to 30 at the RP2D of STI-7349 alone to conduct an expansion study of STI-7349 alone to further assess the safety and preliminary efficacy of the RP2D of STI-7349 alone. STI-7349 will be administered at the same frequency as that in Part 1A and continued until the maximum 2-year dosing period, disease progression/relapse, death, intolerable toxicity, inability of the subject to benefit from study treatment as judged by the investigator, withdrawal from clinical study treatment by the subject or his/her legal representative, loss to follow-up, or completion of the entire study, whichever comes first.

Period II: Dose escalation for STI-7349 in combination with Pembrolizumab (2A) Periond 2A1 part: According to the single-agent RP2D of STI-7349 determined in phase I, the dose of STI-7349 combined with palibrizumab was increased in subjects with advanced solid tumors. ≤ ½RP2D of STI-7349 single agent was used as the starting dose of the combined dose increase, and the expected RP2D dose was 4.8mg. The initial dose of combined administration was ≤2.4mg. The approved standard therapeutic dose of pabolizumab is 200mg IV. According to the results of the Phase I study, the three dose groups of STI-7349 combined with pabolizumab were initially set as 1mg, 1.6mg and 2.4mg, respectively. Qualified subjects will be selected into 3 dose groups in sequence from low to high dose.

Periond 2A2 part: According to the single-agent RP2D of STI-7349 determined in phase I, the dose of STI-7349 combined with other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) was increased in subjects with advanced solid tumors. 1mg (≤ ½RP2D of STI-7349 single agent) was used as the starting dose of the combined dose increase. The investigator will refer to the CSCO or other current guidelines or appropriate drug inserts to determine the dose and dosing schedule of other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.). According to the results of the Phase I study, the two dose groups of STI-7349 combined with other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) were initially set as 1mg, 1.6mg, respectively. Qualified subjects will be selected into 2 dose groups in sequence from low to high dose.

Period II: Dose expansion for STI-7349 in combination with Pembrolizumab (2B) Periond 2B1 part: According to the data from the 2A1 escalation period, target tumor types with potential benefit are selected, and subjects are expanded to 20 to 30 at the RP2D of the combination to conduct a dose expansion study of STI-7349 in combination with Pembrolizumab or add standard treatment on the basis of STI-7349 combined with pembrolizumab to further assess the safety and preliminary efficacy of the RP2D of the combination. STI-7349 will be administered at the same frequency as that in Part 2A1 and continued until the maximum 2-year dosing period, disease progression/relapse, death, intolerable toxicity, inability of the subject to benefit from study treatment as judged by the investigator, withdrawal from clinical study treatment by the subject or his/her legal representative, loss to follow-up, or completion of the entire study, whichever comes first.

Periond 2B2 part：According to the data from the 2A2 escalation period, target tumor types with potential benefit are selected, and subjects are expanded to 20 to 30 at the RP2D of the combination to conduct a dose expansion study of STI-7349 in combination with with other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) or add standard treatment on the basis of STI-7349 combined with with other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) to further assess the safety and preliminary efficacy of the RP2D of the combination. STI-7349 will be administered at the same frequency as that in Part 2A2 and continued until the maximum 2-year dosing period, disease progression/relapse, death, intolerable toxicity, inability of the subject to benefit from study treatment as judged by the investigator, withdrawal from clinical study treatment by the subject or his/her legal representative, loss to follow-up, or completion of the entire study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

-

To be enrolled in this study, subjects must meet all of the following inclusion criteria:

1. Subjects should have fully understood the study and voluntarily signed an informed consent form.
2. Age 18 to 80 years (inclusive).
3. ECOG(Eastern U.S. Oncology Collaborative Group) score of 0 to 1.
4. Expected survival ≥ 12 weeks.
5. According to Response Evaluation Criteria in Solid Tumors (RECIST1.1), the subject has at least one measurable lesion, that is, the subject has at least one lymph node lesion (minimum diameter ≥ 1.5 cm) or non-lymph node lesion (maximum diameter ≥ 1 cm) diagnosed by computed tomography (CT)/magnetic resonance imaging (MRI) examination; if the lesion that previously received local therapy (radiotherapy, ablation, vascular intervention, etc.) is the only lesion, there must be a clear imaging basis for disease progression of this lesion after local therapy.
6. Subjects with malignant advanced solid tumors confirmed by histopathology or cytology who have failed standard treatment, or cannot tolerate standard treatment, or cannot obtain standard treatment for various reasons, or have no standard treatment.
7. The subject has major organ function meeting the following criteria within 7 days prior to first dose [The subject had not received blood component transfusion within 14 days prior to testing. Subjects had not received supportive treatment with human granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), thrombopoietin receptor agonist, interleukin-11, and erythropoietin (EPO) within 7 days prior to testing.]:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   2. Platelet (PLT) ≥ 100 × 109/L;
   3. Hemoglobin (HGB) ≥ 90 g/L;
   4. Alanine aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN(Upper limit of normal value) if liver involvement is known);
   5. Aspartate aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN if liver involvement is known);
   6. Total bilirubin (TBIL) ≤ 1.5 × ULN (≤ 3.0 × ULN if Gilbert's syndrome is diagnosed);
   7. Serum creatinine ≤ 1.5 × ULN or estimated glomerular filtration rate (eGFR, calculated according to the Cockcroft-Gault formula, or by measuring 24-hour urine) ≥ 40 mL/min;
   8. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
8. The toxic reaction of previous anti-tumor therapy returned to ≤ grade 1 (except for the following cases: Grade 2 neurotoxicity and grade 2 hypothyroidism caused by anti-tumor therapy, hair loss and pigmentation of any grade, grade 2 AE that cannot be returned to ≤ grade 1 and will remain stable for a long time as determined by the investigator based on the actual clinical situation, laboratory detection indicators are shown in inclusion Criterion 7) .
9. Subject is willing and able to comply with the study schedule and all other study protocol requirements.
10. Women of childbearing potential (women of non-childbearing potential are defined as sexually mature women who have undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy or bilateral tubal ligation/occlusion, or who are unable to have children because of congenital or acquired disease, or have natural menopause for ≥ 12 months) must have a negative blood pregnancy test during screening. Female subjects of childbearing potential and male subjects must use a highly effective method of contraception at screening through 6 months after the last treatment.

Exclusion Criteria:

-

To be enrolled in this study, subjects must not meet any of the following exclusion criteria:

1. The subject has a known hypersensitivity to any component of the investigational product or IL-2.
2. Subjects have participated in any therapeutic clinical study within 28 days prior to first dose, were enrolled and treated. In addition, subjects are in the survival follow-up phase of observational or interventional studies.
3. Subjects have used immunomodulatory drugs within 14 days or 5 half-lives (whichever is longer) prior to the first dose, including but not limited to thymosin, IL-2, IL-15, interferon, etc.
4. The subject has received chimeric antigen receptor T-cell immunotherapy (CAR-T) within 3 months prior to the first dose; the subject has received chemotherapy (at least 6 weeks for chemotherapeutic agents nitrosoureas and mitomycin C, and at least 14 days for oral fluoropyrimidines), endocrine therapy, targeted therapy (washout period of 14 days or 5 half-lives for small-molecule targeted therapy, whichever is longer), immunotherapy (for immunomodulatory agents see exclusion criterion 3), tumor embolization, etc. within 28 days prior to the first dose; the subject has received radiotherapy within 14 days prior to the first dose, palliative radiotherapy for symptom control is allowed to be completed at least 7 days prior to the first dose; the subject has received traditional Chinese medicine for an approved indication of anti-tumor within 7 days prior to the first dose.Except when subjects assessed by the investigator could be enrolled.
5. The subject has undergone major surgery within 28 days or minor surgery within 7 days prior to the first dose, or had an unhealed wound, ulcer, or bone fracture or required elective surgery during the study (except for diagnostic biopsy, insertion of vascular access device).
6. Subjects have received a live attenuated vaccine within 28 days prior to the first dose or plan to receive it during the study.
7. Subjects have received systemic immunosuppressants within 28 days prior to first dose excluding:

   1. Intranasal inhaled topical steroid therapy or topical steroid injection (eg, intra-articular injection);
   2. Systemic corticosteroid therapy not exceeding 10 mg/day prednisone or its physiologic equivalent doses;
   3. Corticosteroids as prophylaxis for allergic reactions (eg, premedication for CT);
   4. As prophylaxis for infusion reactions.
   5. See exclusion criteria 8 for systemic use of sex hormones in patients with brain metastases.
8. Active central nervous system (CNS) metastases or cancerous meningitis with known or symptomatic symptoms at the screening stage (Note: ① Patients with CNS metastases with symptoms prior to initial administration who have been treated and stable for ≥4 weeks and have been off systemic sex hormone therapy (at any dose) for >3 days may be included. ②Asymptomatic brain metastases (i.e. no neurological symptoms, no need for corticosteroids, and no lesions >1.5cm) can be enrolled, but regular brain imaging examinations are required as a disease site).
9. Subjects had uncontrolled third space effusions requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (subjects who do not require drainage of effusion or have no significant increase in effusion after stopping drainage for 3 days may be enrolled), or third space effusions that are bloody by diagnostic puncture.
10. The subject had another malignancy within 5 years prior to the first dose, except for radically treated early malignancies (carcinoma in situ or Stage I tumor), such as adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast after radical resection, early papillary thyroid carcinoma, or prostate cancer with local Gleason score ≤ 6.
11. The subject had active autoimmune or inflammatory diseases, including inflammatory bowel disease (eg, ulcerative colitis or Crohn's disease), diverticulitis (other than diverticular disease), celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome or Wegener' s syndrome (granuloma with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.), or a history of the disease within the previous 2 years (subject with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic therapy within the last 2 years, hypothyroidism requiring thyroid hormone replacement therapy only, and Type 1 diabetes mellitus requiring insulin replacement therapy only may be enrolled).
12. The subject has active or uncontrolled HBV（Hepatitis B Virus） (HBsAg positive and/or HBcAb positive and HBV DNA titer positive), HCV (HCV-Ab positive and HCV RNA titer positive), HIV(Human Immunodeficiency Virus) positive.
13. The subject had an active bacterial, viral, or fungal infection (defined as a subject demonstrating persistent signs/symptoms related to infection that do not improve despite appropriate antibiotic or other therapy) or required intravenous (IV) antibiotics within 72 hours prior to the first dose.
14. Severe or uncontrolled cardiovascular or cerebrovascular disease requiring treatment, including but not limited to:

    1. New York Heart Association (NYHA) cardiac functional classification > 2;
    2. Unstable angina not controlled by medication;
    3. Subject has had a myocardial infarction within 6 months prior to first dose;
    4. History of myocarditis;
    5. Cardiac tamponade;
    6. Poorly controlled arrhythmias (eg, subjects who develop ventricular tachycardia during antiarrhythmic drug therapy will be excluded; subjects with first degree atrioventricular block or asymptomatic left anterior bundle branch block/right bundle branch block will not be excluded);
    7. 12-lead electrocardiogram QTcF（The QT interval values were corrected for heart rate using Fridericia's formula） > 470 msec;
    8. Left ventricular ejection fraction (LVEF) < 50%;
    9. Poorly controlled hypertension (On the basis of lifestyle modification, the subject has been taking adequate doses of 2 or more antihypertensive agents reasonably tolerated for more than 1 month, but blood pressure remains substandard. Or subjects have been taking 4 or more antihypertensive drugs for effective blood pressure control) or hypotension;
    10. Epilepsy not controlled by medication;
    11. The subject had a stroke, cerebrovascular accident, or transient ischemic attack within 6 months prior to first dose.
15. The subject has known chronic obstructive pulmonary disease (COPD) and forced expiratory volume in one second (FEV1) < 50% of predicted normal. It should be noted that subjects suspected of having COPD must have FEV1 testing and must be excluded if FEV1 is < 50% of predicted normal.
16. The subject has known moderate or severe persistent asthma, or had a history of asthma within the past 2 years, or has uncontrolled asthma of any classification currently (note that subjects with current controllable intermittent asthma or controllable mild persistent asthma are allowed).
17. The subject has previous and current pulmonary disease such as interstitial pneumonia (including drug-induced), pneumoconiosis, pulmonary fibrosis, or severely impaired pulmonary function; the subject has active pulmonary tuberculosis and is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within 1 year prior to the first dose.
18. The subject has experienced clinically significant bleeding symptoms within 3 months prior to first dose. The subject had evident symptoms of coughing up blood within 28 days prior to the first dose with hemoptysis of half a teaspoon (2.5 mL) or more per session.
19. The subject had a history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to the first dose.
20. The subject had a history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism (except thrombosis caused by a vascular access device, or superficial venous thrombosis) within 3 months prior to the first dose.
21. The subject has hepatic encephalopathy, or hepatorenal syndrome, or Child-Pugh class B (> 7 points) or more severe cirrhosis.
22. The subject had a known history of primary immunodeficiency.
23. The subject had a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation (except corneal transplantation).
24. Pregnant or lactating women.
25. Subject has any active serious psychiatric disorder, medical condition, or other symptoms/conditions that could affect treatment, compliance, or ability to give informed consent at the discretion of the investigator.

    The following exclusion criteria apply only to combined dosing subjects:
26. Previous allergy to pabolizumab or other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.).
27. Permanent discontinuation of drug related AE due to pabolizumab or other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) or similar drugs.
28. Permanent discontinuation of the drug due to previous allergy to standard treatment or occurrence of drug-related AE.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants of STI-7349 alone with treatment-related adverse events as assessed by CTCAE v5.0. | Up to 2 years.
  Assessing the incidence of adverse events (AEs) of STI-7349 alone using the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0)
Number of participants of STI-7349 in combination with Pembrolizumab or other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) with treatment-related adverse events as assessed by CTCAE v5.0. | Up to 2 years.
  Assessing the incidence of adverse events (AEs) of STI-7349 in combination with Pembrolizumab or other approved PD-1/PD-L1 inhibitors (e.g., Tislelizumab, etc.) using the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0)

SECONDARY OUTCOMES:
To assess the AUC(Area under the concentration-time curve) of cationic lipids of STl-7349 alone in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the pharmacokinetics(PK) of cationic lipids of STl-7349 alone by collecting serum at protocol-specified time points:AUC.
To assess the Tmax(Time to peak) of cationic lipids of STl-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of cationic lipids of STl-7349 alone by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax(Peak concentration) of cationic lipids of STl-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of cationic lipids of STl-7349 alone by collecting serum at protocol-specified time points:Cmax.
To assess the AUC of mRNA(messenger-ribonucleic acid) of STl-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STl-7349 alone by collecting serum at protocol-specified time points:AUC.
To assess the Tmax of mRNA of STl-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STl-7349 alone by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax of mRNA of STI-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STl-7349 alone by collecting serum at protocol-specified time points:Cmax.
To assess the AUC of HSA-IL2v protein(Human serum albumin interleukin 2 fusion protein) of STl-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STl-7349 alone by collecting serum at protocol-specified time points:AUC.
To assess the Tmax of HSA-IL2v protein of STI-7349 alone in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STl-7349 alone by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax of HSA-IL2v protein of STI-7349 alone in the treatment of advanced solid tumors. | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STl-7349 alone by collecting serum at protocol-specified time points:Cmax.
To assess the AUC of cationic lipids of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of cationic lipids of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:AUC.
To assess the Tmax of cationic lipids of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of cationic lipids of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax of cationic lipids of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of cationic lipids of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Cmax.
To assess the AUC of mRNA of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:AUC.
To assess the Tmax of mRNA of ST1-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax of mRNA of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of mRNA of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Cmax.
To assess the AUC of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:AUC.
To assess the Tmax of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Tmax.
To assess the Cmax of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | The first four cycles(each cycle is 21 days).
  To assess the PK of HSA-IL2v protein of STI-7349 in combination with Pembrolizumab by collecting serum at protocol-specified time points:Cmax.
To assess the ORR(Objective response rate) of STl-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects with CR(Complete Response)+PR(Partial Response) for the best response assessed according to the RECIST 1.1 criteria.
To assess the DCR(Disease control rate) of STI-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects whose best response was CR+PR+SD(Stable Disease) as assessed according to RECIST 1.1 criteria.
To assess the DOR(Duration of response) of STl-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the first onset of CR or PR and the onset of PD(Progressive Disease) or death from any cause (whichever occurs first).
To assess the PFS(Progression-free survival) of STl-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the subject's initial study treatment and the onset of PD or death from any cause, whichever occurs first.
To assess the OS(Overall survival)of STl-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between a subject's initial study treatment and death from any cause.
To assess the the ORR of STl-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects with CR+PR for the best response assessed according to the RECIST 1.1 criteria.
To assess the DCR of STl-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects whose best response was CR+PR+SD as assessed according to RECIST 1.1 criteria.
To assess the DOR of STl-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the first onset of CR or PR and the onset of PD or death from any cause (whichever occurs first).
To assess the PFS of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the subject's initial study treatment and the onset of PD or death from any cause, whichever occurs first.
To assess the OS of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between a subject's initial study treatment and death from any cause.
To assess the anti-PEG(polyethylene glycol) ADA(immunogenicity) of STI-7349 alone in the treatment of advanced solid tumor. | Through study completion, an average of 2 years.
  Change from baseline in anti-PEG ADA contents measured in plasma and correlation with PK/PD(pharmacodynamics).ADA blood sample collection time point:Within 1 week before injection, each cycle before administration(each cycle is 21 days) and at EOT(End-of-treatment visit).
To assess the anti-HSA-IL2v ADA content of STI-7349 alone in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Change from baseline in anti-HSA-IL2v ADA contents measured in plasma and correlation with PK/PD.ADA blood sample collection time point:Within 1 week before injection, each cycle before administration(each cycle is 21 days) and at EOT.
To assess the anti-PEG ADA of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Change from baseline in anti-PEG ADA contents measured in plasma and correlation with PK/PD.ADA blood sample collection time point:Within 1 week before injection, each cycle before administration(each cycle is 21 days) and at EOT.
To assess the anti-HSA-IL2v ADA of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Change from baseline in anti-HSA-IL2v ADA contents measured in plasma and correlation with PK/PD.ADA blood sample collection time point:Within 1 week before injection, each cycle before administration(each cycle is 21 days) and at EOT.
To assess the anti-Pembrolizumab Nab of STI-7349 in combination with Pembrolizumab in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Change from baseline in anti-Pembrolizumab Nab contents measured in plasma and correlation with PK/PD.ADA blood sample collection time point:Within 1 week before injection, each cycle before administration(each cycle is 21 days) and at EOT.
To evaluate the safety, tolerability, and efficacy of STI-7349 in combination with pembrolizumab plus standard therapy in subjects with advanced solid tumors | Up to 2 years.
  Assessing the incidence of adverse events (AEs) of STI-7349 in combination with pembrolizumab plus standard therapy in subjects using the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0)
To assess the the ORR of STI-7349 in combination with pembrolizumab plus standard therapy in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects with CR+PR for the best response assessed according to the RECIST 1.1 criteria.
To assess the DCR of STI-7349 in combination with pembrolizumab plus standard therapy in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the proportion of subjects whose best response was CR+PR+SD as assessed according to RECIST 1.1 criteria.
To assess the DOR of STI-7349 in combination with pembrolizumab plus standard therapy in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the first onset of CR or PR and the onset of PD or death from any cause (whichever occurs first).
To assess the PFS of STI-7349 in combination with pembrolizumab plus standard therapy in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between the subject's initial study treatment and the onset of PD or death from any cause, whichever occurs first.
To assess the OS of STI-7349 in combination with pembrolizumab plus standard therapy in the treatment of advanced solid tumors | Through study completion, an average of 2 years.
  Defined as the time between a subject's initial study treatment and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, Doctor(M.D.), Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine., Yiwu, Zhejiang, China